CLINICAL TRIAL: NCT07071428
Title: A Randomized Controlled Trial on the Treatment of Chronic Tic Disorder With Nourishing the Vital Energy and Regulating the Spirit Needle Technique
Brief Title: Acupuncture Treatment in Pediatric Patients With Tic Disorders: A Prospective, Single-Center, Randomized Controlled Trial
Acronym: ATPTD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Hong Gao, Deputy dean, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ZSLL-ZN-2021-008-01
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Tic Disorders
Keywords: conventional treatment; acupuncture; pediatric; clinical trial; Tic Disorders
MeSH Terms: conditions — Tic Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- therapy group (Experimental)
  Interventions: Procedure: the Nourishing the vital energyand Regulating the spirit needle technique
- control group (Active Comparator)
  Interventions: Procedure: Regular acupuncture

INTERVENTIONS:
Procedure: Regular acupuncture — Primary acupoints: Baihui (GV20), Hegu (LI4, bilateral), Fengchi (GB20, bilateral), Taichong (LV3, bilateral), Jinsuo (GV8), and Ganshu (BL18, bilateral). Operational procedures: Preoperative preparation identical to the treatment group; for Baihui (GV20), perform subcutaneous insertion backward (0.5 cun); for Fengchi (GB20), apply oblique insertion toward the nasal tip (0.8 cun); for Hegu (LI4) and Taichong (LV3), use perpendicular insertion (0.5 cun); for back-shu points (Ganshu BL18), rapid needling is applied due to low safety and inconvenience of retaining needles. Needle manipulation for qi activation, cycle, and frequency align with the treatment group. Treatment protocol: 3 sessions per week, 10 sessions constituting one course, totaling 20 sessions.
  Arms: control group
Procedure: the Nourishing the vital energyand Regulating the spirit needle technique — Primary points: Zhongwan (RN12), Xiawan (RN10), Qihai (RN6), Guanyuan (RN4), Taixi (KI3/bilat.), Baihui (GV20), Sishencong (EX-HN1), Shenting (GV24), Benshen (GB13/bilat.). Supplemental points: Blinking: Zanzhu (BL2) + Taiyang (EX-HN5/affected); Mouth twitch: Dicang (ST4) + Jiache (ST6/affected); Neck twitch: Fengchi (GB20) + Shangqu (KI17/affected); Limb twitch: UL-Waiguan (SJ5) + Quchi (LI11/affected), LL-Futu (ST32) + Yanglingquan (GB34/affected); Vocal tics: Tongue Three Needles (HN23). Post-disinfection: Calm child pre-needling. Sequence: Scalp → abdomen → limbs. Techniques: Scalp points-subcutaneous backward 0.5in; Taixi (KI3)-perpendicular 0.5in, mild lift-thrust/twirl to deqi; Abdomen-abdominal acupuncture (linea alba ref.), adipose/fascial layer insertion (no muscle/deqi), 30min retention no manipulation; Rapid withdrawal with pressure. Protocol: 3 sessions/week, 10-session course, 20 sessions total.
  Arms: therapy group

SUMMARY:
This study was conducted to observe the efficacy of Nourishing the vital energy and Regulating the spirit needle technique in the treatment of chronic tic disorder through the Yale Global Tic Severity Scale (YGTSS) and the Chinese Medicine Symptom Rating Scale in order to provide a new, safe and feasible treatment option and idea for the treatment of chronic Tic Disorder.

DETAILED DESCRIPTION:
In this study, 76 children who met the diagnostic criteria for chronic tic disorder were collected and randomly divided into the therapy group(n-38)and control group(n=38) according to a random number table. The patients were treated 3 times a week for 7 weeks, a total of 20 times. YGTSS scores and the Chinese Medicine Symptom Rating Scale were performed before and after 2 courses of treatment, and clinical efficacy and adverse events were observed in both groups, and YGTSS scores were recorded at follow-up 4 week safter the end of treatment and 12 weeks after the end of treatment, respectively. All data were statistically processed and analysed using SPSS 25.0 software, and relevant differences were compared after processing and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with tic disorders per the Diagnostic and Statistical Manual of Mental Disorders, version 5 (DSM-5) criteria Presence of either motor tics or vocal tics with symptoms present for at least 3 months Aged 5-18 years (all genders) No tic-related medications or therapies for 8 weeks before treatment Willing to complete 8-week acupuncture treatment

Exclusion Criteria:

* Secondary tics from structural neurological lesions (e.g., epilepsy), pharmacologically induced tics, or neurodevelopmental comorbidities Severe communication barriers or cognitive impairments affecting trial participation Severe organ dysfunction meeting clinical diagnostic thresholds Concurrent participation in interventional clinical trials History of acupuncture-related syncope or presyncope episodes Absolute contraindications to acupuncture (e.g., severe needle phobia, skin infections at acupoints)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
The Yale Global Tic Severity Scale | at baseline (pre-treatment), after 8-week treatment, after 4-week follow-up
  The Yale Global Tic Severity Scale (YGTSS) Score is designed to assess the severity of symptoms in children with Tourette's Syndrome by scoring the type of tics, frequency of tics, intensity of tics, complexity of tics, degree of interference with normal behavior, and degree of impairment of social functioning in the child, with a total score ranging from 0-75, with higher scores indicating greater severity of the child's condition.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Gao, Principal Investigator — Third Affiliated Hospital of Zhejiang Chinese Medical University
Locations (1):
- the Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No